CLINICAL TRIAL: NCT03958591
Title: Effects of Short-Term Intensive De-escalation Therapy on Long-term Regimen Simplification in Patients With Poorly Controlled Type 2 Diabetes-- a Multicenter, Open-labeled, Randomized Controlled Trial
Brief Title: Effects of Short-term Intensive De-escalation Therapy on Long-term Regimen Simplification
Acronym: ESTIMATOR
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yanbing Li (Other)
Responsible Party: Sponsor-Investigator, Yanbing Li, Professor, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018YFC1314103
Record Dates: First submitted 2019-05-20; First posted 2019-05-22 (Actual); Last update posted 2022-04-08 (Actual); Status verified 2022-03

CONDITIONS: Diabetes type2
Keywords: poorly controlled diabetes; intensive insulin therapy; wearable device
MeSH Terms: interventions — Wearable Electronic Devices

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intensive-de-escalation group with intelligent management (Experimental): Short-term continuous subcutaneous insulin infusion and thereafter the combination therapy of basal insulin, metformin and vildagliptin will be applied. Then the oral hypoglycemic therapies will be prescribed. Wearable devices and smart apps will be used to manage and follow-up patients.
  Interventions: Drug: CSII and thereafter combination therapy, followed up with wearable devices
- Intensive-de-escalation group without intelligent management (Experimental): Short-term continuous subcutaneous insulin infusion and thereafter the combination therapy of basal insulin, metformin and vildagliptin will be applied. Then the oral hypoglycemic therapies will be prescribed. Traditional ways such as telephone contact will be used to follow-up patients.
  Interventions: Drug: CSII and thereafter combination therapy, followed up in traditional ways
- Traditionally upgrading group (Active Comparator): The combination therapy of basal insulin, metformin and vildagliptin for the entire 12 weeks and thereafter the oral hypoglycemic therapies will be applied. Traditional ways will be used to follow-up patients.
  Interventions: Drug: Traditionally upgrading therapy, followed up in traditional ways

INTERVENTIONS:
Drug: CSII and thereafter combination therapy, followed up with wearable devices — Short-term continuous subcutaneous insulin infusion and thereafter the combination therapy of basal insulin, metformin and vildagliptin; Wearable devices and smart apps will be used to manage and follow-up the participants.
  Other Names: Intensive intelligence group
  Arms: Intensive-de-escalation group with intelligent management
Drug: CSII and thereafter combination therapy, followed up in traditional ways — Short-term continuous subcutaneous insulin infusion and thereafter the combination therapy of basal insulin, metformin and vildagliptin; Traditional ways such as telephone contact will be used for follow up.
  Other Names: Intensive group
  Arms: Intensive-de-escalation group without intelligent management
Drug: Traditionally upgrading therapy, followed up in traditional ways — The participants will be applied the combination therapy of basal insulin, metformin and vildagliptin for the entire 12 weeks. Traditional ways will be used for follow up.
  Other Names: Traditional group
  Arms: Traditionally upgrading group

SUMMARY:
Despite advances in diabetes management, many patients with type 2 diabetes in China fail to achieve optimal glycemic control. One of the possible reasons is associated with the delay in therapeutic decision making that lags behind glycemic rise. The investigators design this study and presume that using vildagliptin and metformin in combination with basal insulin as sequential treatment after intensive insulin therapy, might better modulate the dual islet hormone dysfunction than traditionally stepwise upgrading therapy pattern in patients with poorly controlled T2DM, and thus lead to a glucose normalization, β-cell function improvement and therapy simplification.

DETAILED DESCRIPTION:
This is a multicenter, randomized, controlled, open-label, clinical superiority trial. The participants will be recruited from 19 centers in China. The enrolled participants will be randomly assigned into 3 groups, designated as Group A , B and C.

Group A (Intensive therapy group following up with intelligent equipment)：Continuous subcutaneous insulin infusion (CSII) will be applied to the participants for 2 weeks and thereafter the combination therapy of basal insulin, metformin and vildagliptin for the next 10 weeks. The participants are followed up with intelligent equipment.

Group B (Intensive therapy group following up in traditional ways): CSII will be applied to the participants for 2 weeks and thereafter the combination therapy of basal insulin, metformin and vildagliptin for the next 10 weeks. The participants are followed up in traditional ways.

Group C (Traditionally upgrading group): The participants will be applied the combination therapy of basal insulin, vildagliptin and metformin for the entire 12 weeks.

Participants in both Group A, B and Group C will then receive combination therapy of metformin and vildagliptin, and be followed-up at the 16th, 20th, 24th, 28th, 32nd and 36th weeks. The doses of metformin and vildagliptin are set as 1.0~2.0g/d and 100mg/d, respectively. If the participants cannot tolerate metformin, then acarbose (50-100mg tid) or SGLT2 inhibitor can be instead used. If glucose is not well controlled, sulfonylureas or glinides can be added as a rescue treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Type 2 diabetes diagnosed according to WHO criteria (1999); With a duration of 1~10 years;
2. With two or more oral hypoglycemic drug used for at least 3 months, including at least one insulin secretagogue in half-max dosage (eg. Glibenclamide 7.5mg/d, gliclazide 60mg/d, glimepiride 3mg/d, glipizide 10mg/d, repaglinide 6mg/d, nateglinide 360mg/d and DPP-4 inhibitor with regular doses);
3. HbA1c of 7.5 to 13% and fasting C-peptide >0.4 nmol/L;
4. Age of 18 to 70 years;
5. BMI of 20 to 35 kg/m²；
6. Capable of and willing to follow doctors' instructions to:

   * Self-monitor blood glucose according to the protocol;

     * Follow the protocol and have regular visits as required; ③ Record and maintain the research diary, as required by the protocol; ④ Keep contact with the investigators and receive phone calls during the study.

Exclusion Criteria:

1. Type 1 diabetes or specific types of diabetes;
2. Those who have received premixed insulin therapy and/or basal - meal insulin and/or basal insulin-oral hypoglycemic agents treatment accumulation for 7 days or more, and those who have received CSII therapy in the last one year, and those who have received GLP-1 analogue within 3 months before screening;
3. Those who have acute diabetic complications (diabetic ketoacidosis, hyperosmotic hyperglycemia coma or lactic acidosis);
4. Those who have severe diabetic microvascular complications (proliferative retinopathy, clinical proteinuria, and glomerular filtration rate less than 45 ml/min, uncontrolled diabetic neuropathy and obvious diabetic autonomic neuropathy);
5. Those with ALT >2.5 times of the upper limit of normal (ULN), bilirubin > 1.5 times of ULN；
6. Those with known macrovascular disease: Patients with acute cerebrovascular accident, acute coronary syndrome, unstable angina, peripheral artery disease who have received vascular intervention or amputation in the 12 months before enrollment; Or chronic cardiac dysfunction with cardiac function grade III or above;
7. Those with poor blood pressure control (systolic blood pressure≥160mmHg and/or sitting diastolic blood pressure ≥110mmHg) and inability to control under 160/110mmhg within 1 week;
8. Serious systemic disease or malignant tumor, chronic diarrhea, etc；
9. Those with drugs that may affect blood glucose for a cumulative time of more than 1 week within 12 weeks, such as oral/venous glucocorticoid, growth hormone, estrogen/ progesterone, high-dose diuretics, antipsychotic drugs. However, low-dose diuretics for antihypertensive purposes (HCTZ < 25mg/d, indapamide < 1.5mg/d) and physiologic dose of thyroid hormone for replacement therapy are not included；
10. Any factors that may affect the participation of the subject in the study or the evaluation of the results；
11. Pregnancy or planned pregnancy, lactation subjects.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 274 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
the proportions of treatment simplification | 24 weeks after the insulin treatment
  the proportions of patients who can maintain glycemic targets (HbA1c<7%) with only combination of oral hypoglycemic agents

CONTACTS AND LOCATIONS:
Overall Officials: Yanbing Li, Dr, Principal Investigator — FAH-SYSU
Locations (1):
- Department of endocrinology, FAH-SYSU, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No